CLINICAL TRIAL: NCT02150213
Title: A Multicenter Medical Safety Follow-up Study for Patients With Partial Onset Seizures Who Received More Than 28 Days of Total Exposure to BGG492 in Studies CBGG492A2207 and/or CBGG492A2212
Brief Title: Medical Safety Follow-up Study for Patients Who Received More Than 28 Days of Total Exposure to BGG492
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CBGG492A2216; 2013-003431-29 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-29 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Adrenocortical Adenoma; Endometrial Stromal Sarcomas
Keywords: Adrenocortical Adenoma,; Endometrial Stromal sarcomas; BGG492
MeSH Terms: conditions — Adrenocortical Adenoma; Sarcoma, Endometrial Stromal | interventions — Magnetic Resonance Spectroscopy; Postmortem Imaging; High-Energy Shock Waves; Biopsy; selurampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BGG492 (Experimental): This was a follow-up safety study where study treatment was not administered. Patients came from BGG492 studies where patients were previously exposed to > 28 days of BGG492 50 mg, 100 mg or 150 mg given orally three times a day
  Interventions: Procedure: MRI, CT or ultrasound was permitted if MRI was contraindicated; Procedure: Dexamethasone Supression Test; Procedure: Sonogram; Procedure: Biopsy; Drug: BGG492

INTERVENTIONS:
Procedure: MRI, CT or ultrasound was permitted if MRI was contraindicated — MRI/CT/ultrasound of abdomen
  Other Names: Magnetic Resonance Imaging Computed tomography
Procedure: Dexamethasone Supression Test — Low dose of dexamethasone is administered in the evening; the next morning, a blood sample is collected to measure cortisol
Procedure: Sonogram — Sonogram of the uterus (females only)
  Other Names: Sonogram ultrasound
Procedure: Biopsy — Uterine endometrial biopsy (females only)
  Other Names: Uterine Biopsy
Drug: BGG492 — No study-drug was administered in this study
  Other Names: Selurampanel

SUMMARY:
To provide medical follow-up to patients exposed to BGG492 for more than 28 days in study CBGG492A2207 (NCT 01147003) and/or CBGG492A2212 (NCT 01338805).

DETAILED DESCRIPTION:
The purpose of the study was to provide medical follow-up to patients exposed to BGG492 for more than 28 days in study CBGG492A2207 (NCT 01147003) and/or CBGG492A2212 (NCT 01338805). Data from study CBGG492A2216 was used to support the clinical safety assessment of BGG492 regarding the observance of uterine endometrial stromal tumors and adrenal cortical adenomas at least one year after the completion of BGG492 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent had to be obtained before any assessment was performed;
2. Patients had to be cooperative, willing to participate in the study assessments, and be able to report AEs (adverse events) themselves or have a caregiver who can record and report the events;
3. Total exposure to BGG492 treatment in Study BGG492A2207 and/or BGG492A2212 had to have been greater than 28 days
4. At least 1 year had to have elapsed since the patient received his or her last dose of BGG492.

Exclusion Criteria:

- There were no exclusion criteria for this study. All patients meeting the inclusion criteria were eligible to participate in the follow-up safety assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (4):
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Hoffman, New Jersey
  - Novartis Investigative Site, Dallas, Texas
- Germany (5):
  - Novartis Investigative Site, Bernau
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Kehl-Kork
  - Novartis Investigative Site, Ulm
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szombathely
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
- Slovakia (3):
  - Novartis Investigative Site, Hlohovec, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica, Slovakia
- Novartis Investigative Site, Seoul, Korea, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of this follow-up safety study was to provide medical follow-up to patients exposed to BGG492 for more than 28 days in Study BGG492A2207 and/or BGG492A2212.
Pre-assignment Details: The first period focused on contacting the patients, obtaining consent for follow-up, and conducting screening assessments. The second period of the study focused on performing the follow-up procedures, obtaining and interpreting the results, and referring the patient, if necessary, to an appropriate medical specialist.
Period: Overall Study
Arm/Group | BGG492
Started | 59
Completed | 57
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Includes all patients who signed the informed consent form for the study.
Arm/Group | BGG492
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (11.58)
Gender [Count of Participants; unit: Participants]
  Female | 31
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adrenal Cortical Adenomas
Description: Incidence of adrenal cortical adenomas as assessed by non-contrast MRI of the abdomen (CT or ultrasound of the abdomen was permitted if MRI was contraindication)
Time Frame: Minimum of one year after last dose of BGG492 in study BGG492A2207 or BGG492A2212
Population: Full analysis Set: included all patients who signed informed consent to enter the study
Measure: Number; unit: Particpants
Arm/Group | BGG492
Number analyzed (Participants) | 59
Particpants | 3

2. Primary Outcome: Incidence of Uterine Endometrial Stromal Sarcomas
Description: Incidence of uterine endometrial stromal sarcomas as assessed by sonogram/biopsy (females)
Time Frame: Minimum of one year after last dose of BGG492 in study BGG492A2207 or BGG492A2212
Population: Full Analysis Set (FAS):included all patients who signed informed consent to enter the study, but this assessment was only done on female patients. Of the 31 female patients, two had a hysterectomy and were not evaluated (N=29)
Measure: Number; unit: Participants
Arm/Group | BGG492
Number analyzed (Participants) | 29
Participants | 0

ADVERSE EVENTS:
Arm/Group | BGG492
Serious Adverse Events (participants affected / at risk) | 5/59
Other Adverse Events (participants affected / at risk) | 3/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BGG492 (N=59)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BGG492 (N=59)
Renal Cyst (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.